CLINICAL TRIAL: NCT02661308
Title: Reducing Cancer Side-effects With Systematic Light Exposure
Acronym: LYS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Ali Amidi, Cand.psych, Ph.D., Aarhus University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Sagsnr. 1-10-72-286-15
Record Dates: First submitted 2015-12-15; First posted 2016-01-22 (Estimated); Last update posted 2024-06-28 (Actual); Status verified 2024-06

CONDITIONS: Cancer-related Fatigue; Cancer-related Cognitive Impairment

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- Systematic bright light exposure (Experimental): Systematic bright light exposure for 30 min. for 4 weeks
  Interventions: Device: Litebook
- Systematic dim light exposure (Active Comparator): Systematic dim light exposure for 30 min. for 4 weeks
  Interventions: Device: Litebook

INTERVENTIONS:
Device: Litebook

SUMMARY:
The main purpose of this interdisciplinary proposal is to conduct two randomized controlled trial (RCT) of the efficacy of self-administered systematic light exposure (Bright White Light (BWL)), an innovative, low cost, and low burden intervention to treat cancer-related fatigue. Another common and often overlapping treatment side-effect is cognitive impairment. A secondary outcome of the proposed RCT is, thus, cognitive functioning. Finally, possible underlying chronobiological (circadian activity rhythms, sleep), biological (pro inflammatory markers), and neurophysiological (brain morphology) mechanisms of BWL will be explored.

DETAILED DESCRIPTION:
Two independent but similar RCTs with a total of 144 breast cancer patients (Group 1 = 72 high risk patients; Group 2 = 72 low risk breast cancer patients) post-treatment screened for fatigue will be randomized to BWL (36 in each of the two groups) or dim light(DL) (36 in each of the two groups) exposure for 30 minutes/morning for 4 weeks, and assessed before, during, immediately and 3 months after the intervention. Measures include questionnaires, cognitive assessment, actigraphy, blood samples, saliva samples, and magnetic resonance imaging (MRI).

1.1 Aims and hypotheses. Aim 1: To test the efficacy of BWL on fatigue (primary outcome) in breast cancer patients.

Hypothesis 1: Compared with control participants exposed to DL, participants randomized to BWL will report less fatigue immediately and 3 months after the intervention.

Aim 2: To test the efficacy of BWL on cognitive functioning (secondary outcome).

Hypothesis 2: Compared with controls, BWL recipients will show improved cognitive functioning immediately and 3 months after the intervention.

Aim 3: To explore the effects of BWL on chronobiological, biological, and neurophysiological markers.

Hypothesis 3: BWL will be associated with normalized circadian activity rhythms (3a); improved sleep (3b); decreased inflammation (3c); increased cortical and subcortical grey matter density (3d); and increased cortical and subcortical white matter integrity (3e). If hypotheses 1 and/or 2 are confirmed, the mediating effects of the markers will be explored.

ELIGIBILITY:
Inclusion Criteria - Group 1:

* High-risk breast cancer patients as defined by the Danish Breast Cancer Cooperative Group (DBCG) having received treatment according to the DBCG guidelines
* Minimum age of 18 years; completion of adjuvant whole breast radiation treatments
* A score <34 on the FACIT-Fatigue scale (see below) after radiotherapy
* Availability for home-based 4-week BWL/DL-treatment.

Exclusion Criteria:

* History of chronic fatigue disorders
* Pregnancy
* Confounding underlying medical illnesses such as significant pre-existing anemia
* Diagnosed or suspected psychiatric or medical condition that might contribute to fatigue (other than those caused by the cancer or its treatment)
* History of bipolar disease or mania (which are contra-indications for light treatment)
* Current clinical depression
* History of seasonal affective disorder
* Previous diagnosis of sleep apnea, restless legs or other sleep disorders (not including insomnia) known to affect fatigue
* Employment in shift work
* Chronic use of oral steroid medication
* Prior use of light treatment
* Use of photosensitising medications
* Plans to travel across meridians
* Insufficient Danish language proficiency

Inclusion criteria - Group 2:

* Low-risk postmenopausal patients as defined by the DBCG having received breast-conserving surgery for lymph node-negative breast cancer
* Completion of adjuvant whole breast radiation treatments
* A score <34 on the FACIT Fatigue scale (see below) after radiotherapy
* Availability for home-based 4-week BWL/DL-treatment.

Exclusion Criteria:

* History of chronic fatigue disorders
* Pregnancy
* Confounding underlying medical illnesses such as significant pre-existing anemia
* Diagnosed or suspected psychiatric or medical condition that might contribute to fatigue (other than those caused by the cancer or its treatment)
* History of bipolar disease or mania (which are contra-indications for light treatment)
* Current clinical depression
* History of seasonal affective disorder
* Previous diagnosis of sleep apnea, restless legs or other sleep disorders (not including insomnia) known to affect fatigue
* Employment in shift work
* Chronic use of oral steroid medication
* Prior use of light treatment
* Use of photosensitising medications
* Plans to travel across meridians
* Insufficient Danish language proficiency

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Cancer-related fatigue (FACIT-fatigue) | Changes in fatigue from baseline to immediately after intervention (T1-T2)
Cancer-related fatigue (FACIT-fatigue) | Changes in fatigue from baseline to 3 months after intervention

SECONDARY OUTCOMES:
Pittsburgh Sleep Quality Index (PSQI) | Immediately after intervention and 3 months after intervention
Beck's Depression Inventory - II (BDI-II) | Immediately after intervention and 3 months after intervention
Connors Continous performance test (CPT-3) | Immediately after intervention
Psychomotor vigilance test (PVT) | Immediately after intervention
Hopkins Verbal Learning Test (HVLT-R) | Immediately after intervention
Health-related quality of life (SF-36) | Immediately after intervention and 3 months after intervention
Anxiety symptoms (HADS Anxiety) | Immediately after intervention and 3 months after intervention
Impact of events (IES-R) | Immediately after intervention and 3 months after intervention
Patients assessment of own functioning Inventory (POAFI) | Immediately after intervention and 3 months after intervention
Overall neuropsychological composite score | Immediately after intervention and 3 months after intervention

OTHER OUTCOMES:
Mediators: Changes in brain white mater diffusion integrity as measured with diffusion-weighted MR imaging: Diffusion/kurtosis parameters. | Immediately after intervention
Mediators: Changes in Pro-inflammatory cytokines (Il-1, Il-6, Tnf-alpha) (blood draw) | Changes from baseline to immediately after intervention
Mediators: Changes in circadian activity rhythms (actigraphy) | Changes from baseline to immediately after intervention
Mediators: Changes in diurnal Cortisol (saliva samples) | From baseline to immediately after intervention
Mediators: Changes in diurnal melatonin (as measured with saliva samples) | From baseline to immediately after intervention
Mediators: Changes in grey matter density as measured by T-1 weighted MR imaging (voxel-based morphometry) | Immediately after intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus Universitets Hospital, Aarhus, Denmark